CLINICAL TRIAL: NCT02522975
Title: A Prospective, Randomized, Double Blind, Parallel Group Study to Establish the Therapeutic Equivalence of EPIAO® With the Standard Treatment EPREX® in Subjects With Chronic Kidney Disease (CKD) Related Anaemia Not Yet on Dialysis
Brief Title: Biosimilar Erythropoietin in Anaemia Treatment (Correction Phase Study)
Acronym: BEAT_001
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Shenyang Sunshine Pharmaceutical Co., LTD. (Industry)
Collaborators: Navitas Life Sciences GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SSS_EP_001
Record Dates: First submitted 2015-08-10; First posted 2015-08-14 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Renal Anaemia
Keywords: biosimilar epoetin; efficacy; safety; immunogenicity; renal anaemia
MeSH Terms: interventions — Epoetin Alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Reference group (Active Comparator): Generic name: recombinant human erythropoetin injection which is indicated for the treatment of anaemia caused by chronic renal disease.
  Dosage form:Injection Strength:2000IU,3000IU,4000IU Frequency and Dosage:subcutaneously injection once a week for a period of 52 weeks. The initial dose of EPREX® will be 60 IU/kg body weight.
  Interventions: Drug: EPREX®
- Experimental group (Experimental): Generic name: recombinant human erythropoetin injection which is indicated for the treatment of anaemia caused by chronic renal disease.
  Dosage form:Injection Strength:2000IU,3000IU,4000IU Frequency and Dosage:subcutaneously injection once a week for a period of 52 weeks. The initial dose of EPIAO® will be 60 IU/kg body weight.
  Interventions: Drug: EPIAO®

INTERVENTIONS:
Drug: EPIAO® — Recombinant human erythropoietin falls under the pharmacological class of haematopoietic / anti anaemic agents. It has been developed for the treatment of anaemia in subjects with chronic kidney disease.
  Erythropoietin, also known as EPO, is a glycoprotein hormone that controls erythropoiesis, or RBC production. It is a cytokine (protein signalling molecule) for erythrocyte precursors in the bone marrow. Human EPO has a molecular weight of 34,000.
  Other Names: Recombinant human erythropoietin
  Arms: Experimental group
Drug: EPREX® — Recombinant human erythropoietin falls under the pharmacological class of haematopoietic /anti anaemic agents. It has been developed for the treatment of anaemia in subjects with chronic kidney disease.
  Erythropoietin, also known as EPO, is a glycoprotein hormone that controls erythropoiesis, or RBC production. It is a cytokine (protein signalling molecule) for erythrocyte precursors in the bone marrow. Human EPO has a molecular weight of 34,000.
  Other Names: Recombinant human erythropoietin
  Arms: Reference group

SUMMARY:
This study is aimed to comprehensively establish the biosimilarity/bioquivalence in EPIAO® and EPREX® in terms of 52-week comparisons in efficacy,safety and immunogenicity.The targeted population is anaemia patients with chronic renal disease who are naive to epoetin treatment and not yet on haemodialysis.

DETAILED DESCRIPTION:
This is a prospective, randomized, double blind, parallel group two arm study to establish the therapeutic equivalence, safety and tolerability of EPIAO® as compared to EPREX® in the treatment of CKD related anaemia in subjects who are not yet on dialysis (pre-dialysis). A total of 96 subjects will be randomized into two groups in a 1:1ratio. Treatment arm A will receive EPIAO® once a week, subcutaneously for period of 52 weeks and treatment arm B will receive EPREX, weight once a week, subcutaneously for period of 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects between the age of 18 to 75 years
2. Subjects with renal anaemia (haemoglobin 7.5 g/dl to 10 g/dl)
3. Subjects who are treatment naïve to epoetin
4. Subjects with chronic kidney disease (CKD) stages* 3 and 4 not yet on dialysis (predialysis)
5. Subjects willing to provide a written informed consent
6. Subjects with serum ferritin ≥ 100 μg/L and/or transferrin saturation ≥ 20%

   * CKD staging will be based on the five-stage system for classification of CKD based on KDIGO guidelines.

Exclusion Criteria:

1. Subjects with anaemia due to other reasons (that is not renal anaemia)
2. Subjects on dialysis
3. Subjects who have undergone blood transfusion within the last 3 months
4. Subjects with major complication such as severe/chronic infections or bleeding, or aluminum toxicity
5. Subjects with suspected or known PRCA
6. Subjects with a history of aplastic anaemia
7. Subjects with uncontrolled diabetes (fasting blood glucose > 240 mg/dl) or uncontrolled hypertension (systolic blood pressure > 180 mm Hg, diastolic blood pressure > 110 mm Hg)
8. Subjects with known hypersensitivity to any of the ingredients of the investigational products, the mammalian cell-derived product or human albumin products
9. Subjects with history of seizure disorder
10. Subjects with hematological disorder (thrombocytopenia, neutropenia, or hemolysis)
11. Subjects with hyperparathyroidism (intact parathyroid hormone > 1000 pg/ml)
12. Subjects with severe liver dysfunction
13. Subjects with congestive heart failure and/or angina (NYHA class III and IV)
14. Subjects with myocardial infarction or stroke in the preceding 6 months of screening
15. Subjects with active malignancy in the previous 5 years
16. Subjects with gastrointestinal bleeding in the past 6 months
17. Subjects with immunosuppressive therapy in the previous 3 months
18. Subjects with Hepatitis B virus (HbsAg), Hepatitis C virus (HCV), Human Immunodeficiency Virus (HIV) and syphilis
19. Female subjects who are pregnant, breast-feeding,planning to be pregnant during the study, or women of child-bearing potential (any woman who is not surgically sterile i.e. bilateral tubal ligation, total hysterectomy or < 2 years post menopause) not using a reliable method of double contraception (e.g. condom plus diaphragm, condom or diaphragm plus spermicidal gel/foam, tubal ligation, or stable dose of hormonal contraception) throughout the study period
20. Subjects participating in trials involving erythropoietin in the past 6 months before screening
21. Subjects currently participating or participation in an investigational study within 30 days prior screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-08; Primary Completion 2019-06 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Mean absolute change in haemoglobin(Hb) | 24 weeks
  Mean absolute change in haemoglobin(Hb) level from baseline to 24 weeks after treatment with EPIAO®/EPREX® in parallel groups (g/dl),respectively."

SECONDARY OUTCOMES:
Mean absolute change in weekly epoetin dosage | 24 weeks
  Mean absolute change in weekly epoetin dosage per kg body weight from baseline to 24 weeks after treatment with EPIAO®/EPREX® in parallel groups (IU/kg/week).
Frequency of adverse events | 52 weeks
  To observe the frequency of adverse events following EPIAO® and EPREX® administration.
Occurence of anti-epoetin antibodies | 52 weeks
  To monitor the occurrence of anti-epoetin antibodies among subjects following at least 52 weeks of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: BOLONG MIAO, Ph.D, Study Director — Shenyang Sunshine Pharmaceutical Co., LTD.
Locations (8):
- Thailand (8):
  - Bamrasnaradura Infectious Disease Institute, Bangkok
  - Bhumibol Adulyadej hospital, Bangkok
  - BMA hospital, Bangkok
  - Chulalongkorn King Memorial hospital, Bangkok
  - Klongton Hospital, Bangkok
  - Phramongkutklao hospital, Bangkok
  - Rajavithi hospital, Bangkok
  - Siriraj Hospital, Bangkok